CLINICAL TRIAL: NCT03778450
Title: Long-term Opioid Therapy, Misuse and Mortality in Patients With Chronic Non-cancer Pain in Germany
Status: Completed | Type: Observational
Sponsor: LinkCare GmbH (Industry)
Collaborators: Grünenthal GmbH (Industry); Klinikum Saarbrücken (Unknown); Ruhr University of Bochum (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Tino Schubert, Managing Partner, LinkCare GmbH
Other Study IDs: VF_1014_1040_Study Protocol
Record Dates: First submitted 2018-12-07; First posted 2018-12-19 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Analgesics, Opioid: Patients are only included if they have been diagnosed in at least three quarters in the study period with one of the following diagnoses: R51, R52*, M00*-M99*, G43*-G44*, G50.0 or G50.1, F45.4*, G62*, or E10.4*-E14.4 plus G63.3. At least one diagnoses must be between 1 January 2012 and index treatment and main and secondary hospital diagnoses (i.e. Haupt- und Nebendiagnosen) will be used to include the patients.
  Interventions: Drug: Analgesics, Opioid
- Non-Opioid Analgesic: Patients are only included if they have been diagnosed in at least three quarters in 2012 with one of the following diagnoses: R51, R52*, M00*-M99*, G43*-G44*, G50.0 or G50.1, F45.4*, G62*, or E10.4*-E14.4 plus G63.3.At least one diagnoses must be between 1 January 2012 and index treatment and main and secondary hospital diagnoses (i.e. Haupt- und Nebendiagnosen) will be used to include the patients.
  Interventions: Drug: Non-Opioid Analgesic

INTERVENTIONS:
Drug: Analgesics, Opioid — Patients are included in the long-term opioid group if they started an opioid-therapy between 2013 and 2017 and received consecutive prescriptions for opioid medications over a minimum of 3 quarters, over a 60-month period between January 1, 2013, and December 31, 2017. The treatment will be assessed using the ATC codes of opioid
  treatment N02AA01, N02AA05, N02AB03, N02AE01, N02AX02, N02AX01, N02AX06) reported in reimbursed medicines to patients.
  Other Names: Opioid Group
  Groups: Analgesics, Opioid
Drug: Non-Opioid Analgesic — Patients with non-opioid pain medication are included, if they received a medication therapy with anticonvulsants (gabapentin, pregabalin, carbamazepine), antidepressants or non-opioid analgesics (NSAIDs, Metamizole) over a minimum of 3 quarters, over a 60-month period between January 1, 2013, and December 31, 2017. The non-opioid treatment will be assessed using the ATC codes (N03AX12, N03AX16, N03AF01) of treatment reported in reimbursed medicines to patients.
  Other Names: Non-Opioid Group
  Groups: Non-Opioid Analgesic

SUMMARY:
Among patients receiving opioids for noncancer pain, recent research in North America showed a strong association between doses and opioid-related mortality, especially at dosages exceeding thresholds recommended in recent guidelines. However, the focus on over-dosage may underestimate overall opioid-related mortality and data on death associated with opioid use in a population-based cohort of chronic noncancer pain patients in Europe is scarce. Especially comparative studies studying the safety of long-term opioid therapy in a real-world setting relative to non-opioid medication for chronic noncancer pain are needed in a European context.

DETAILED DESCRIPTION:
This is a cross-sectional observational cohort study between 2012 and 2017 of patients with chronic noncancer pain. The primary objective is to investigate the association between mortality among patients with chronic noncancer pain with long-term opioid-therapy compared to non-opioid pain medication. The data will be retrieved from an anonymized German health claims database including 4,00,000 persons insured by 69 German statutory health insurances. The data set includes 5.0% of the population covered by statutory health insurances from January 1, 2012, to December 31, 2017. Only anonymized and aggregated data (no directly or indirectly identifying data) will be extracted.

Patients with headache, diseases of the musculoskeletal system and connective tissue, migraine, trigeminal neuralgia, atypical facial pain, persistent somatoform pain disorder, polyneuropathies, or diabetes mellitus with neurological complications in at least 3 quarters between 01.01.2012 and their first pain medication claim are analyzed. Patients will be stratified in an opioid and a non-opioid group and will be compared with a propensity score matching approach.

Patients' follow-up period include 5 years after start treatment and chronic pain diagnosis between 01.01.2013 and 31.12.2017. Each patient will be censored at death (death date), switching of study group, 12 months without treatment or followed-up 5 years until last known record for the, whichever happens first. The main analyses will be analyzed with a multivariate Cox proportional hazards regression.

ELIGIBILITY:
Inclusion Criteria:

- Patients are only included if they have been diagnosed in at least three quarters in the study period with one of the following diagnoses: R51, R52*, M00*-M99*, G43*-G44*, G50.0 or G50.1, F45.4*, G62*, or E10.4*-E14.4 plus G63.3. At least one diagnoses must be between 1 January 2012 and index treatment and main and secondary hospital diagnoses (i.e. Haupt- und Nebendiagnosen) will be used to include the patients.

Exclusion Criteria:

* Patients with present opioid and non-opioid pain medication prescriptions in 2012 are excluded from analysis (therapy-naïve patients only).
* Cancer patients will be excluded if the cancer diagnosis is accompanied by at least one of the following treatments in the same quarter: radiation therapy or chemotherapy all defined by the OPS codes in. Diagnoses will be assessed via ICD-10 diagnoses during the inclusion period from 1 January 2012 until index treatment and main and secondary hospital diagnoses (i.e. Haupt- und Nebendiagnosen) will be taken into account.
* Palliative care, coded by ICD-10 code Z51.5 or OPS code 8-982*, 8-98e*, 8-98h* before index date is excluded
* Opioid substitution treatment with ICD-10 code Z51.83 in the study period is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The database contains data on around 4 million insured people from 69 German statutory health insurances (SHI). German SHI system comprises of approximately 120 independent health insurance companies. Funds paid by these SHI to any provider of health care (e.g. hospitals, physicians, pharmacies, psychotherapists and physiotherapists) represent almost the complete picture of the total health care costs of individual patients. All health insurance data can be linked to patients' demographics including age and gender. T
Sampling Method: Non-Probability Sample
Enrollment: 3232 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 2013 - 2017
  Primary endpoint is death by any course in the study follow-up. Death will be assessed during the follow-up period by number of patients who deceased during follow-up period (2013 - 2017) via the date of death in German claims data base.

SECONDARY OUTCOMES:
Hospitalization due to any course | 2013 - 2017
  Hospitalization will be assessed via the number of hospitalisations (calculated by counting the number of discharge dates (KH_Fall. Entlassungsdatum) in the year of interest, hospitalization rate. The rate of hospitalization will be estimated as the number of patients with at least one hospitalization during the follow-up period divided by person-time of follow-up, censoring at time of death, last known record for the patient in the database, or 31st December 2017 (end of latest data cut), whichever is earlier.
Number of ICU-stays | 2013 - 2017
  Intensive care unit (ICU-stay) stay is defined as patient's stay based on specialty of departement in hospital (KH_OPS.Fachabteilung = 3600).
Hospitalization with to misuse or addiction | 2013 - 2017
  The hospitalization with misuse or addiction will be analysed, if principal (main) diagnosis at discharge date between January 1st 2013 and December 31st 2017 contains at least one ICD-10 diagnosis of misuse/addiction: F10* or F11* or F13* or F19* or T40*
Number of coding of procedures in hospitals | 2013 - 2017
  Coding of procedures in hospitals that indicate number of patients that were hospitalized with severe diseases such as cardiovascular diseases will be assessed via OPS-Codes provided in the protocol
Number of patients with a ca misuse or addiction diagnosis in the outpatient sector | 2013 - 2017
  The number of patients with a least one coding of ICD 10 codes of a misuse or addiction diagnosis in the outpatient sector will be assessed via number of codings of misuse/addiction (ICD Codes = F10* or F11* or F13* or F19* or T40*) in outpatient sector by general practitioner or a specialist (e.g. psychiatrist), as ensured diagnosis (Diagnosesicherheit='G').
Number of sick leave days | 2013 - 2017
  Sick leave will be assessed as an absolute number number of days being off work of patients in 2013-2017 .
Number of hospital deaths | 2013 - 2017
  Hospital deaths will be assessed via reason of discharge = death (Entlassgrund = Tod)
Number of main- and secondary discharge diagnoses | 2013 - 2017
  Main- and secondary discharge diagnoses from hospital deaths will be assessed as the TOP 20 diagnoses of patients who deceased during a hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Tino Schubert, Study Director — LinkCare GmbH
Locations (1):
- LinkCare GmbH, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauser W, Schubert T, Vogelmann T, Maier C, Fitzcharles MA, Tolle T. All-cause mortality in patients with long-term opioid therapy compared with non-opioid analgesics for chronic non-cancer pain: a database study. BMC Med. 2020 Jul 15;18(1):162. doi: 10.1186/s12916-020-01644-4. PMID 32664901

DOCUMENTS (1):
  • Study Protocol (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03778450/Prot_000.pdf